CLINICAL TRIAL: NCT05918679
Title: Improving Speech Motor Learning Processes Using Augmented Behavioral Interventions
Brief Title: The Brain Processes Underlying Speech Motor Learning and Speech Production
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00017657; R01DC019905 (NIH)
Record Dates: First submitted 2023-06-05; First posted 2023-06-26 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Healthy Adults group 1 (Experimental)
  Interventions: Behavioral: Effects of speech variability on speech motor learning
- Healthy Adults group 2 (Experimental)
  Interventions: Behavioral: Effects of error-detection training on speech motor learning
- Healthy Adults group 3 (Experimental)
  Interventions: Behavioral: Contributions of error awareness to speech motor learning
- Healthy Adults group 4 (Experimental)
  Interventions: Behavioral: Enhancing auditory-to-motor mapping with augmented visual feedback
- Healthy Adults group 5 (Experimental)
  Interventions: Behavioral: Effects of enhanced auditory-motor awareness on speech motor learning

INTERVENTIONS:
Behavioral: Effects of speech variability on speech motor learning — This intervention will examine whether reducing normal variability of speech could improve error detection and speech motor learning. We will design training tasks to change subjects' speech variability. We will train subjects to decrease/decrease their speech variability. Upon completing the training tasks, subjects will complete a motor learning task.
  Arms: Healthy Adults group 1
Behavioral: Effects of error-detection training on speech motor learning — This intervention will examine whether improving subjects' ability to detect and estimate auditory perturbation could improve speech motor learning. For this purpose, we will design training tasks to change subjects' estimation of the perturbation magnitude. After completing the training tasks, subjects will complete the motor learning task.
  Arms: Healthy Adults group 2
Behavioral: Contributions of error awareness to speech motor learning — This intervention will examine the contributions of error awareness to speech motor learning. Subjects will produce a target word while receiving perturbed auditory feedback with different magnitudes. Subjects will be trained to indicate the magnitude of the error they perceived with or without visual feedback.
  Arms: Healthy Adults group 3
Behavioral: Enhancing auditory-to-motor mapping with augmented visual feedback — This intervention will determine the contributions of enhanced auditory-to-motor mappings to speech motor learning. We will design training tasks in which we will use visual feedback to provide feedback regarding subjects' accuracy of auditory-to-motor mapping.
  Arms: Healthy Adults group 4
Behavioral: Effects of enhanced auditory-motor awareness on speech motor learning — In this intervention, subjects will be trained to control their articulators more accurately and be more aware of their articulators' position and their auditory consequences. After the training tasks, subjects will complete a motor learning task.
  Arms: Healthy Adults group 5

SUMMARY:
The aim of this research is to develop protocols that selectively target and improve speech-motor learning processes. Participants will be asked to name pictures, read words/sentences, and listen to sounds while their speech signals will be collected during the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* native speaker of American English
* normal (age-appropriate) binaural pure-tone hearing threshold
* not taking medications affecting sensorimotor functioning
* no current or history of communication, neurological, or psychological disorders

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in speech output in response to previously experienced auditory errors | within each session of the study that may last up to 2 hours
  In each trial, participants will experience an auditory error while they produce speech (e.g., they may say "head" but hear "had"). Participants' speech will be measured in each trial. The investigators will measure how the participants' speech changes due to auditory errors experienced in previous trials.
Change In Speech Output Immidiately After Hearing Auditory Errors | within each session of the study that may last up to 2 hours
  In each trial, participants will experience an auditory error while they produce speech (e.g., they may say "head" but hear "had"). The investigators will measure how the participants' speech changes due to auditory errors that they experience in the current trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Tempe, Arizona, United States